CLINICAL TRIAL: NCT03759405
Title: Myocardial Cell Vein Transplantation for Chronic Heart Failure
Brief Title: IPS Differentiated Cardiomyocytes Vein Transplantation for Chronic Heart Failure
Acronym: IDCVTCHF
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing University of Chinese Medicine (Other)
Collaborators: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Anlong Xu, professor, Beijing University of Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUCM
Record Dates: First submitted 2018-11-23; First posted 2018-11-30 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic heart failure treatment group (Experimental): One case of CHF caused by coronary heart disease, one case of CHF caused by dilated heart disease and one case of CHF caused by Keshan disease were selected and treated with autologous iPS differentiated cardiomyocyte intravenous transplantation.
  Interventions: Biological: iPS differentiated cardiomyocytes

INTERVENTIONS:
Biological: iPS differentiated cardiomyocytes — Repair of injured myocardium by vein transplantation with autologous iPS differentiated cardiomyocytes

SUMMARY:
Based on the safety evaluation of primates, the best cell transplantation scheme was integrated. One patient with CHF caused by coronary heart disease, one patient with CHF caused by dilatation and one patient with CHF caused by Keshan disease were selected and treated with autologous iPS differentiated cardiomyocyte intravenous transplantation. The safety evaluation of human body was completed and combined with subjective and objective indexes respectively. Structural and functional indicators were used to evaluate the therapeutic effect of cell transplantation. The results of animal experiments confirmed the safety and effectiveness of intravenous myocardial cell transplantation, and clarified its possible mechanism.

ELIGIBILITY:
Inclusion Criteria:

* It accords with the diagnostic standard of chronic heart failure.
* The etiological diagnosis accords with the corresponding diagnostic standard.
* The age is 30~80 years old.
* Cardiac function classification is III- grade IV.
* Signed informed consent.

Exclusion Criteria:

* Those who did not meet the diagnostic criteria and were included in the standard.
* Patients with severe dyspnea (such as COPD with pulmonary encephalopathy, upper gastrointestinal bleeding, etc.) accompanied by obvious hypoxemia and hemodynamic instability.
* Patients with severe primary diseases, such as liver and kidney diseases, hematological diseases, autoimmune diseases, malignant tumors, progressive diseases or diseases with poor prognosis, such as severe infection, severe water and electrolyte disorders, acid-base imbalance.
* Various infectious diseases.
* Participants in other clinical trials in the past two months.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2022-12-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessment | 6 months
  Minnesota Heart Failure Scale for Quality of Life. Scale ranges (0-100), do higher values represent a worse outcome. The higher the score, the lower the quality of life.
Curative effect evaluation | 6 months
  Cardiac Function Measurement by Cardiac Color Doppler Ultrasound. Under normal conditions, left ventricular ejection fraction is more than 50%. The lower ejection fraction, the worse heart function.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No